CLINICAL TRIAL: NCT07161843
Title: Determine the Efficacy of Investigational Drug QRX-3 in Hospitalized Patients With Acute Tubular Necrosis Pattern of Acute Renal Failure
Brief Title: Use of QRX-3 for Acute Tubular Necrosis Type of Renal Failure in Hospitalized Patients ( QRX-3 in ARF)
Acronym: QRX-3 in ARF
Status: Not yet recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Ebima Clifford Okundaye (Industry)
Responsible Party: Sponsor-Investigator, Ebima Clifford Okundaye, President, Neukidney Inc.
Organization: Neukidney Inc. (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 0002
Record Dates: First submitted 2025-04-10; First posted 2025-09-09 (Actual); Last update posted 2025-09-09 (Actual); Status verified 2025-09

CONDITIONS: Acute Renal Failure (ARF); Acute Tubular Necrosis
Keywords: acute renal failure; acute tubular necrosis
MeSH Terms: conditions — Acute Kidney Injury; Kidney Cortex Necrosis

STUDY DESIGN:
Intervention Model Description: added QRX-3 to standard regime
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Use of QRX-3 in addition to standard therapy (Experimental): QRX-3 drug orally as twice daily in addition to standard conventional therapy will be given to this group for 28 days
  Interventions: Drug: QRX-3
- control group (Placebo Comparator): placebo twice daily will be given to this group in addition to standard therapy
  Interventions: Drug: QRX-3

INTERVENTIONS:
Drug: QRX-3 — Combination of QRX-3 with standard therapy will be given to one arm in trial , another arm will receive placebo
  Other Names: Eseronate

SUMMARY:
Use of QRX-3 in hospitalized patients with pediatric and adult patients with acute tubular necrosis renal failure

ELIGIBILITY:
Inclusion Criteria:

* Hospitalized patients
* presence of Acute renal failure
* Nephrologist diagnosis of Acute tubular necrosis or fractional excretion of sodium of >2%
* willingness to participate

Exclusion Criteria:

High risk of bleeding Absence of hydronephrosis or obstructive uropathy Absence of baseline dialysis use single kidney status

Ages: 10 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 500 (Estimated)
Dates: Start 2025-08-30 (Estimated); Primary Completion 2026-12-30 (Estimated); Study Completion 2027-02-01 (Estimated)

PRIMARY OUTCOMES:
Rate of change in creatinine glomerular filtration rate | 28 days
  compare the outcome effect of added QRX-3 drug to placebo in addition to standard therapy on the rate of change from baseline of creatinine GFR in ATN patients

SECONDARY OUTCOMES:
daily change in glomerular filtration rate in ml/min | 7 days
  daily change in GFR by creatinine in mls/min
daily change in cystatin C level in mg/dl | 7 days
  daily change in measured cystatin C level

OTHER OUTCOMES:
effect of QRX-3 on recovery of renal function in patients with ATN renal failure | 28
  comparism of number of patient achieving return to baseline renal function in both groups

CONTACTS AND LOCATIONS:
Locations (1):
- Neukidney Inc, Rosharon, Texas, United States

IPD SHARING:
Plan to Share IPD: Undecided